CLINICAL TRIAL: NCT07273201
Title: Effect of Isolated Versus Synergetic Muscle Facilitation on Upper Limb Functional Performance in Patients With Acute Stroke
Brief Title: Isolated Versus Synergetic Muscle Facilitation on Upper Limb Functional Performance in Acute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed Mousa, Assistant lecturer of physical therapy for neurology and neurosurgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005625
Record Dates: First submitted 2025-11-15; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Acute Stroke
Keywords: acute stroke, upper limb functional performance, muscle facilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- isolated muscle facilitation training (Experimental): Participants in this group will receive a standard physical therapy program including range of motion exercise, electrical muscle stimulation, and Mental practice with motor imagery and stretching exercise, isolated muscle facilitation using electromyography (EMG) biofeedback for six weeks, followed by task-oriented training ofthe upper limb for six weeks
  Interventions: Other: standard physical therapy program; Other: isolated muscle facilitation
- synergistic muscle facilitation training (Active Comparator): Participants in this group will receive a standard physical therapy program, including a range of motion exercise, electrical muscle stimulation, Mental practice with motor imagery, and stretching exercise, synergetic muscle facilitation for six weeks, and followed by task-oriented training of the upper limb for six weeks
  Interventions: Other: standard physical therapy program; Other: synergetic muscle facilitation program

INTERVENTIONS:
Other: standard physical therapy program — * Soft tissue technique (stretch) will be applied for the anterior pectoral region, elbow flexors, pronators, wrist flexors, and finger flexors(for both research groups.
  * Passive Range of motion exercises will be applied for the glenohumeral joint, scapulothoracic articulation, elbow joint, radioulnar joint, and wrist joint(for both research groups).
  * Muscular electrical stimulation will be applied for supraspinatus, anterior and posterior deltoid, biceps and triceps, pronators and supinators, wrist and finger extensors, and finally the lumbricals (Each muscle group 20 min) (for both research groups).
  In mental practice, the patient adheres to a set of imagined task performances ( picking up a cup) or movements (reaching out with the arm).
Other: isolated muscle facilitation — Muscle facilitation exercises will be applied for the anterior deltoid, middle deltoid, posterior deltoid, biceps, triceps, radioulnar pronators and supinators, wrist and finger extensors, wrist and finger flexors, and lumbricals using EMG biofeedback.
  During EMG biofeedback training, the electrodes will be placed on (pectoralis major, triceps, and finger flexor muscles, and (trapezius, biceps, and wrist flexors) to ensure the isolated firing of each muscle group (100 reps each muscle group). Before training, patients should be instructed how to perform muscle contraction exercises according to the displayed EMG signal through multimedia publicity, to improve their coordination. During training, patients can take a sitting or lying down position. Then, the electrode piece will be attached to the abdominal part of the patients' deltoid muscle, triceps brachii, a forearm muscle group, thus collecting the EMG signal generated by the relaxation of the patients' upper limb muscles
  Arms: isolated muscle facilitation training
Other: synergetic muscle facilitation program — Muscle facilitation exercises will be applied for the anterior deltoid, middle deltoid, posterior deltoid, biceps, triceps, radioulnar pronators and supinators, wrist and finger extensors, wrist and finger flexors, and lumbricals During the synergetic muscle facilitation, we will permit the muscles that are linked together through flexion or extension synergy to fire together (100 reps each muscle group) using EMG biofeedback training.
  Arms: synergistic muscle facilitation training

SUMMARY:
This study is a randomized controlled clinical trial that will be carried out to investigate the effect of isolated versus synergetic muscle facilitation on upper limb functional performance in patients with acute stroke.

RESEARCH QUESTION:

Is there a difference between isolated and synergetic muscle facilitation on upper limb functional performance in patients with acute stroke?

It will be hypothesized that:

There will be no difference between isolated and synergetic muscle facilitation on upper limb task-oriented training in patients with acute stroke.

Treatment procedures:

Study group (A): patients will receive a physical therapy program in the form of a range of motion exercise, electrical muscle stimulation, stretching exercise, mental practice with motor imagery, and isolated muscle facilitation using electromyography (EMG) biofeedback for six weeks and followed by task-oriented training of the upper limb for six weeks control group (B): will receive a standard physical therapy program including range of motion exercise, electrical muscle stimulation, Mental practice with motor imagery and stretching exercise, synergetic muscle facilitation for six weeks, and followed by task-oriented training of the upper limb for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral Middle cerebral artery (MCA) stroke patients
* Brunnstrom stage of recovery 1& 2
* Normal body mass index (18.5 - 24.99 kg/m2)
* Dominant handedness

Exclusion Criteria:

* Perceptual, apraxia, major cognitive deficits
* Recurrent stroke
* Subjects with cerebellar lesions, painful or subluxated shoulder, any contracture or deformity of the upper extremity

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of upper limb functional performance (dexterity- coordination) using the Action Reach Arm Test (ARAT) | before enrollment and the end of treatment at 6 weeks
  - Action Reach Arm Test (ARAT): It will be used to assess upper extremity performance (coordination, dexterity, and functioning). It is a 19-item observational measure. Items are categorized into four subscales (grasp, grip, pinch, and gross movement) and arranged in order of decreasing difficulty. Subjects are first asked to perform the most difficult task within a subscale, followed by the least difficult task. while scoring the individual based on their performance of each task
  -Required Equipment: Chair without armrests, Table, Wooden blocks of various sizes, Cricket ball, Sharpening stone, Alloy tubes, Washer and bolt, 2 glasses Sharpening stone, Marbles, Ball bearings, and a Tin lid.
  -scoring: Task performance is rated on a 4-point scale, ranging from 0 (no movement) to 3 (movement performed normally). Scores on the ARAT may range from 0 to 57 points, with a maximum score of 57 indicating better performance.

SECONDARY OUTCOMES:
Analysis of upper limb kinematics (shoulder, elbow, and wrist Positions and acceleration speed of movement) using Kinovea software | Before enrollment and at the end of treatment at 6 weeks
  Kinovea is a valid, precise, and reliable computer program for measuring angles and distances. Kinovia software will be used to analyze the kinematics (Position and acceleration speed)of the shoulder, elbow, and wrist. while patients perform the subscales of the Action Reach Arm Test.
  * Instrumentation: Digital video camera and Computer equipment for the measurement process.
  * procedure: All participants were instructed to wear light clothes for the determination of the selected bony landmarks and to allow easy forward reaching motion. An adhesive marker dot will be placed on preselected anatomical landmarks like the acromion, lateral epicondyle, and wrist (ulnar styloid/mid-forearm) to measure joint angles (shoulder, elbow, wrist) and movement speed. Then, patients will be asked to perform the subscales of the Action Reach Arm Test, such as reaching and grasping. Patients will be captured while performing these tasks using video camera and will be analyzed using Kinovia program.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of Physical Therapy, Cairo University, and El kasr El-Einy hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided